CLINICAL TRIAL: NCT00001844
Title: Functional and Metabolic Imaging Using Magnetic Resonance at 3.0 Tesla
Brief Title: Study of New Magnetic Resonance Methods
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990163; 99-CC-0163
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-09-07

CONDITIONS: Healthy
Keywords: MRI/MRS; Functional MRI; Metabolic Imaging; Brain; Healthy Volunteer

SUMMARY:
This study will evaluate new magnetic resonance imaging (MRI ) methods using a MRI machine more powerful than those in most hospitals. MRI is a diagnostic tool that uses a large magnet and radio waves to produce images of the human body. It can also provide information about brain chemistry and physiology. This study will use the new MRI hardware and methods to measure blood flow and metabolism in regions of the brain during simple tasks, such as listening to tones or watching flashing checkerboards.

Healthy normal volunteers will undergo MRI scanning. For this procedure, the person lies on a stretcher that is moved into a MRI machine, which produces a strong magnetic field. A special lightweight coil is placed on the person's head to obtain better pictures. The scan time ranges from 20 minutes to 2 hours, with the average scan lasting between 45 and 90 minutes.

During the MRI, the person may be asked to perform simple tasks, such as listening to tones or watching a screen, tapping fingers or moving a hand. More complex tasks may require thinking about tones or pictures and responding to them by pressing buttons.

The images produced in this study will be compared with those produced using standard MRI. The results will be used to develop improved imaging methods for better patient care and research.

DETAILED DESCRIPTION:
Technical advances in Magnetic Resonance Imaging (MRI) and Magnetic Resonance Spectroscopy (MRS) has provided researchers with the opportunity to study functional and metabolic changes of the central nervous system (CNS) in both healthy controls and individuals with neurological diseases in response to sensory, motor or cognitive stimulation. While MRI is in common usage in radiology departments and clinics MRI and MRS techniques and hardware are continually being upgraded and designed for Functional Magnetic Resonance Imaging (fMRI) and Magnetic Resonance Spectroscopic Imaging of the CNS at 3.0 Tesla. We will evaluate new sequences on volunteers and for potential use in patients with CNS pathology. These studies are required in order to develop and implement new imaging techniques for research and clinical applications.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. age 18 and older
  2. capable of providing own informed consent
  3. capable of filling out MRI screening form

EXCLUSION CRITERIA:

1. contraindications for MRI including aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body (e.g. metal shavings); or insulin pump, or other metal in the body.
2. pregnancy
3. Subjects will be excluded if it is deemed that they have a condition that would preclude their participation for technical development (e.g. claustrophobia)
4. Subjects will be excluded if they present unnecessary risk (e.g. Brain surgery of uncertain type, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 1999-09-08; Study Completion 2012-09-07

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Frank, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ogawa S, Lee TM, Kay AR, Tank DW. Brain magnetic resonance imaging with contrast dependent on blood oxygenation. Proc Natl Acad Sci U S A. 1990 Dec;87(24):9868-72. doi: 10.1073/pnas.87.24.9868. PMID 2124706
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.
- [Background] Turner R, Howseman A, Rees GE, Josephs O, Friston K. Functional magnetic resonance imaging of the human brain: data acquisition and analysis. Exp Brain Res. 1998 Nov;123(1-2):5-12. doi: 10.1007/s002210050538. PMID 9835386